CLINICAL TRIAL: NCT06202131
Title: Prospective Single-center Study About the Use of Ctdna in the Management of Patients With Tumors of the Gastrointestinal Tract
Brief Title: Use of Ctdna in Patients With Gastrointestinal Tract Tumors
Acronym: ctdna-GI
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6151
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pancreas Cancer; Colon Cancer; Biliary Tract Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Colonic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma ctdna
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate the use of ctDNA in the clinical management of patients with tumors of the gastrointestinal tract.

DETAILED DESCRIPTION:
This is a a prospective observational single-center study; it is a spontaneous study, not sponsored by pharmaceutical companies, and does not involve the use of experimental drugs. The study involves a collection of data, carried out while protecting the anonymity and personal information of individual patients suffering from neoplasms of the gastrointestinal tract, the execution of peripheral blood samples and the collection of faecal material at pre-determined times -points. Circulating biomarkers (as ctDNA) will be evaluated in these samples, in order to optimize both the diagnostic and therapeutic processes of patients with tumors of the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* PS ECOG <2;
* Histological diagnosis of gastrointestinal cancer: esophageal, gastric, intestinal, pancreatic, biliary tract neoplasms;
* Radiological evidence of resectable/locally advanced/metastatic disease on the date of signing the written informed consent;
* Adequate organ and function;
* Availability of tumor histological material.

Exclusion Criteria:

* No histological diagnosis of neoplasia of the gastrointestinal tract.
* No written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old with an histological diagnosis of gastrointestinal tract cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
mOS | 3 years
  The primary endpoint of the study is to evaluate the probability of overall survival (mOS) in relation to the expression of specific molecular markers present in the plasma/faeces of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Sakvatore, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Policlinico Agostino Gemelli, Rome, Lazio, Italy